CLINICAL TRIAL: NCT00823589
Title: Immune Status of Elderly Population Admitted in an Acute Geriatric Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2008 -21
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Aging
Keywords: ELDERLY POPULATION
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pathological group (Experimental): pathological group
  Interventions: Other: Blood test and clinical test
- healthy aged (Experimental): healthy aged
  Interventions: Other: Blood test and clinical test

INTERVENTIONS:
Other: Blood test and clinical test — Blood test and clinical test

SUMMARY:
Ageing is associated with vulnerability against infections leading to increased morbidity with risk of death. Innate and adaptive immunities are altered with ageing responsible of deficits in immune response against pathogens and after vaccination, and favouring the elderly vulnerability against a new pathogen with increased bacterial, viral, and fungal infections.

If immunity has been widely studied in immunosenescence, there are few prospective, comparative studies with elderly ill patients. Moreover among these studies, pathologies are not well defined.

The main objective of our project is to compare the immune state of elderly hospitalised subjects in an acute geriatric unit to the immune state of elderly healthy subjects selected with strict criteria, in order to precise the impact of polypathology and of various pathologies on immunity state.

ELIGIBILITY:
Inclusion Criteria:

* Subject of 75 or more years old, female or male
* Subject admitted in the service of short stay gériatrique of the hospital Holy Marguerite, whatever is the motive for admittance
* Subject not being under supervision(guardianship), nor guardianship
* Subject benefiting from a benefit system
* Subject having given its assent of participation or for which the reliable person gave her assent in the case of vulnerable person

Exclusion Criteria:

* Subject of less than 75 years old
* Subject refusing to participate in the study or for whom(which) the reliable person refuses the participation of the subject

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2009-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
compare the immune state of elderly hospitalised subjects in an acute geriatric unit to the immune state of elderly healthy subjects | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: ELODIE CRETEL, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- HOPITAL DE SAINTE MARGUERITE Service de Gériatrie Sud, Marseille, Paca, France